CLINICAL TRIAL: NCT01446679
Title: Special Drug Use-Results Survey of Lipitor Tablets
Acronym: ALWAYS
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: LIP003
Record Dates: First submitted 2011-09-22; First posted 2011-10-05 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Hypercholesterolemia
Keywords: Lipitor; HMG-CoA reductase inhibitor
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- atrovastatin group: Who receive atrovastatin
  Interventions: Drug: atrovastatin

INTERVENTIONS:
Drug: atrovastatin — oral
  Other Names: Lipitor

SUMMARY:
This study is to evaluate the controlling effect of atrovastatin on plasma lipid to achieve the category-specific targeted lipid levels.

DETAILED DESCRIPTION:
To confirm the low-density lipoprotein cholesterol (LDL-C)-lowering effect of 24 weeks of treatment with Lipitor®(Generic Name : atorvastatin calcium) Tablets and determine the rate of achievement of the category-specific target LDL-C level in patients with hypercholesterolemia; and to confirm the usefulness (efficacy and safety) of atorvastatin in patients who have not responded sufficiently to other statin therapies

ELIGIBILITY:
Patients with hypercholesterolemia who have not achieved the category-specific target lipid level

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hypercholesterolemia who have not achieved the category-specific target lipid level in other statin therapies
Sampling Method: Non-Probability Sample
Enrollment: 24050 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in plasma LDL-C concentration | 0, 4, 12 and 24 week
Change in rate of achievement of the category-specific target LDL-C level | 0, 4, 12 and 24 week

SECONDARY OUTCOMES:
Change in plasma lipid values (LDL cholesterol, HDL cholesterol, triglycerides, total cholesterol, and malondialdehyde-modified LDL [MDL-LDL]) | 0, 4, 12 and 24 week
Changes in renal function test values (urinary albumin, urinary creatinine, urinary protein, and serum creatinine) | 0, 4, 12 and 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contract, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku